CLINICAL TRIAL: NCT00907790
Title: Nursing Management of IBS:Improving Outcomes
Brief Title: Nursing Management of Irritable Bowel Syndrome (IBS) 2008
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Monica Jarrett, Professor, Co-PI, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32722; 2R01NR004142 (NIH)
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Cognitive Therapy; Abdominal Pain; Quality of Life
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive Self-Management (CSM) (Experimental): Comprehensive Self-Management includes 8 sessions that cover education, diet, relaxation training, and cognitive behavioral strategies as they related to symptoms of IBS
  --------------------------------------------------------------------------------
  Interventions: Behavioral: Comprehensive Self-Management (CSM)
- Usual Care (Control Group) (Other): Includes the usual care provided by the person and their health care provider.
  Interventions: Behavioral: Usual Care (Control Group)

INTERVENTIONS:
Behavioral: Usual Care (Control Group)
  Arms: Usual Care (Control Group)
Behavioral: Comprehensive Self-Management (CSM) — Comprehensive Self-Management includes 8 sessions that cover education, diet, relaxation training, and cognitive behavioral strategies as they related to symptoms of IBS
  Arms: Comprehensive Self-Management (CSM)

SUMMARY:
The aim of this study is test the efficacy of a comprehensive self-management therapy to decrease abdominal pain/discomfort and improve quality of life in patients with irritable bowel syndrome (IBS) compared to IBS patients receiving their usual care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women must be: 18-70 years old, have had symptoms of Irritable Bowel Syndrome (IBS) at least 6 mo prior to their diagnosis, and have had their diagnosis for at least 6 months, and the diagnosis had to be made by a health care provider (e.g., internist, gastroenterologist, family, nurse practitioner, physician assistant).
* In addition, the subjects must be experiencing IBS symptoms as described in the Rome-III criteria.161 That is recurrent abdominal pain or discomfort at least 3 days a mo in the last 3 mo associated with 2 or more of the following: improvement with defecation, onset associated with a change in frequency or form (appearance) of their stool.
* Adults 50 or older must have a negative colonoscopy, sigmoidoscopy, abdominal ultrasonography, or barium enema.
* Anyone with a "red flag" symptom (e.g., lost 10 lbs without trying, blood in stool, anemia) will be contacted for additional clarification.

Exclusion Criteria:

* Participants will be excluded if they are taking the following medications: antibiotics, daily use of anticholinergics, tricyclic antidepressants, calcium-channel blockers
* Have a medical history of abdominal surgery (except appendectomy, Caesarian section, tubal ligation, laparoscopic cholecystectomy, hysterectomy, or abdominal wall hernia repair)
* Active organic GI disease, gluten intolerance (celiac disease), or chronic moderate to severe pain condition (e.g., low back pain, fibromyalgia)
* Recent travel to regions with endemic parasitic diseases
* Current mental health disorders (psychosis, bipolar disorder, current moderate to severe depressive episode, suicide attempt, drug or alcohol abuse or dependence within 2yrs)
* Cardiac valvular disease, immune compromised immunologic disorders (e.g., autoimmune conditions)
* Women who are pregnant, breast feeding, or planning to get pregnant in the next year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Daily abdominal pain | Baseline, three and six months post randomization
IBS Quality of Life Questionnaire | Baseline, three and six months post randomization

SECONDARY OUTCOMES:
Salivary cortisol | Baseline, three and six months post randomization
Interleukin-10(IL-10) and Interleukin-12(IL-12) | Baseline, three and six months post randomization
Fecal calprotectin | Baseline, three and six months post randomization
Intestinal permeability (urine) | Baseline, three and six months post randomization
Brief Symptom Inventory | Baseline, three and six months post randomization
Cognitive Scale for Functional Bowel Disorders | Baseline three and six months post randomization
Work Productivity & Activity Impairment | Baseline, three and six months post rand
Daily symptoms(other GI and psychological) | Baseline, three and six months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Maargaret M Heitkemper, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Yang PL, Burr RL, Buchanan DT, Pike KC, Kamp KJ, Heitkemper MM. Indirect effect of sleep on abdominal pain through daytime dysfunction in adults with irritable bowel syndrome. J Clin Sleep Med. 2020 Oct 15;16(10):1701-1710. doi: 10.5664/jcsm.8658. PMID 32620184
- [Derived] Kamp KJ, Weaver KR, Sherwin LB, Barney P, Hwang SK, Yang PL, Burr RL, Cain KC, Heitkemper MM. Effects of a comprehensive self-management intervention on extraintestinal symptoms among patients with IBS. J Psychosom Res. 2019 Nov;126:109821. doi: 10.1016/j.jpsychores.2019.109821. Epub 2019 Aug 29. PMID 31499231
- [Derived] Han CJ, Kohen R, Jun S, Jarrett ME, Cain KC, Burr R, Heitkemper MM. COMT Val158Met Polymorphism and Symptom Improvement Following a Cognitively Focused Intervention for Irritable Bowel Syndrome. Nurs Res. 2017 Mar/Apr;66(2):75-84. doi: 10.1097/NNR.0000000000000199. PMID 28252569